CLINICAL TRIAL: NCT02805530
Title: Radical Treatment of Synchronous Oligometastatic Disease and Primary Tumor in Advanced Non-small Cell Lung Carcinoma (NSCLC)
Brief Title: Radical Treatment of Synchronous Oligometastatic Non-Small Cell Lung Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Medical Sciences Researcher (SNI III), Instituto Nacional de Cancerologia de Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 015/023/ICI
Record Dates: First submitted 2016-05-23; First posted 2016-06-20 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Synchronous Neoplasms
Keywords: oligometastatic disease, radical treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms, Multiple Primary | interventions — Radiotherapy; Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: First line systemic treatment Epidermal growth factor receptor (EGFR)-mutated with tyrosine kinase inhibitors (afatinib, erlotinib or gefitinib). Patients without driver mutation duplet of chemotherapy based on platin taking account histologic subtype (Carboplatin or Cisplatin plus pemetrexed for adenocarcinomas, gemcitabine for epidermoid or paclitaxel for both) at discretion of the treating physician.
  Radical treatment to the primary and to the metastases will be with surgery, radiotherapy, chemoradiotherapy, stereotactic radiosurgery or radiofrequency ablation.
  Radiation: radiation therapy Patients will receive dose and fraction regimen according to the metastatic site.
  Chemoradiotherapy Chemoradiotherapy with duplet based on platins (Carboplatin or cisplatin plus pemetrexed or paclitaxel or etoposide or vinorelbine) or monotherapy with carboplatin.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): Patients with synchronous metastases at Central Nervous System (CNS), evaluated in less than one week by the Multidisciplinary Committee at National Cancer Institute of Mexico to define the initial treatment. Patients with metastases at other sites than CNS will receive first line systemic treatment, in those EGFR-mutated with tyrosine kinase inhibitors (TKI) and in patients without a driver mutation with first line duplet of chemotherapy based on platin. The type of TKI or chemotherapy will be at discretion of the treating physician.
  After 4 cycles of treatment, patients with stable disease or partial response will be evaluated by de Multidisciplinary Committee to establish the type of radical treatment to the primary and to the metastases, radiation therapy and chemoradiotherapy.
  Interventions: Other: First line systemic treatment; Other: Radical treatment; Radiation: radiation therapy; Other: Chemoradiotherapy

INTERVENTIONS:
Other: First line systemic treatment — Epidermal growth factor receptor (EGFR)-mutated with tyrosine kinase inhibitors (afatinib, erlotinib or gefitinib). Patients without driver mutation duplet of chemotherapy based on platin taking account histologic subtype (Carboplatin or Cisplatin plus pemetrexed for adenocarcinomas, gemcitabine for epidermoid or paclitaxel for both) at discretion of the treating physician.
Other: Radical treatment — to the primary and to the metastases will be with surgery, radiotherapy, chemoradiotherapy, stereotactic radiosurgery or radiofrequency ablation.
Radiation: radiation therapy — Patients will receive dose and fraction regimen according to the metastatic site.
Other: Chemoradiotherapy — Chemoradiotherapy with duplet based on platins (Carboplatin or cisplatin plus pemetrexed or paclitaxel or etoposide or vinorelbine) or monotherapy with carboplatin.

SUMMARY:
Non-small cell lung cancer (NSCLC) is the most frequent neoplasm worldwide and also represents the main cause of cancer death. However, it represents the main cause of death by cancer. The prognosis of survival at 5 years is poor, approximately 13-15%.

Various studies suggest that patients who clinically present with a limited number of metastases, a term defined as oligometastatic disease, could have a better prognosis of survival with a radical treatment, than for their counterparts with a greater number of metastasis.

The purpose of this study is to add more information to the current medical literature about the benefits in overall survival of radical treatment of oligometastatic disease in patients with NSCLC and equal or less than 5 synchronous metastases at the time of diagnosis.

The outcomes of the study are to determine the global survival and progression-free survival in patients with synchronous oligometastatic (equal to or less than 5 sites) advanced NSCLC undergoing radical treatment of all metastatic sites and the primary tumor.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is the most frequent neoplasm worldwide and also represents the main cause of cancer death. However, it represents the main cause of death by cancer. The prognosis of survival at 5 years is poor, approximately 13-15%.

The timely detection of NSCLC is difficult and the options for curative treatment are limited since the majority of patients are diagnosed in advanced stages. The standard treatment in metastatic disease is cytotoxic chemotherapy with platins (cisplatin or carboplatin) in combination with a third generation drug (vinorelbine, paclitaxel, docetaxel, gemcitabine or pemetrexed). This therapeutic scheme results in response rates between 20-30%, with a mean overall survival between 8-11 months.

In recent years, research in oncology has focused on the development of therapies aimed at molecular targets that control the growth and proliferation of the tumor cell. Various monoclonal antibodies (bevacizumab, cetuximab) and tyrosine kinase inhibitors (erlotinib, gefitinib, afatinib, crizotinib) have been evaluated with this purpose in NSCLC treatment. Clinical studies in advanced NSCLC, using these new drugs with or without chemotherapy, have had favorable results by increasing the progression-free survival and the response rate, without being able to demonstrate to date, a significant improvement in the overall survival.

Various studies suggest that patients who clinically present with a limited number of metastases, a term defined as oligometastatic disease, could have a better prognosis of survival with a radical treatment, than for their counterparts with a greater number of metastasis.

Much of the current medical information on clinical outcomes in oligometastatic disease is based on clinical studies and retrospective case series of institutions. The majority of the reports have included a mix of patients with synchronous and metachronous oligometastatic disease, focusing on the radical treatment of specific sites such as the brain and adrenal glands. These results have been recognized by the European Society for Medical Oncology (ESMO) and have been included in its treatment guidelines for lung cancer (2012). The recommendation states to consider some radical treatment in selected patients with solitary metastases.

There is limited information about the clinical benefits in overall survival in the subgroup of patients with NSCLC that clinically present with synchronous oligometastatic disease and equal to or less than 5 synchronous metastases at the time of diagnosis.

The purpose of this study is to add more information to the current medical literature about the benefits in overall survival of radical treatment of oligometastatic disease in patients with NSCLC and equal to or less than 5 synchronous metastases at the time of diagnosis. The outcomes of the study are to determine the global survival and progression-free survival in patients with synchronous oligometastatic (equal to or less than 5 sites) advanced NSCLC undergoing radical treatment of all metastatic sites and the primary tumor.

ELIGIBILITY:
Inclusion Criteria:

* Pathology diagnosis of non-small cell lung cancer
* Any histology type (adenocarcinoma, epidermoid carcinoma or large cell carcinoma)
* age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) score 0-1
* Clinical stage IV according to staging system American Joint Committee on Cancer (AJCC) seventh EDITION
* Oligometastatic disease defined as metastases equal to or less than 5 sites.
* Synchronous metastases defined as those that are identified within the first month of the diagnosis of the primary tumor.
* Laboratory results: plasma leukocyte ≥3,000/mm3, platelets ≥100,000/mm3, hemoglobin ≥ 10 gr/dl, serum Creatinine ≤ 1.5 mg/dl, total bilirubin ≤1.5, transaminases ≤ 2.5 times the upper limit of normal (ULN), alkaline phosphatase < 5 times the ULN.
* Candidate to platinum-based chemotherapy.
* Life expectancy estimated with treatment of at least 24 weeks.
* Must have understood and signed the informed consent

Exclusion Criteria:

* Concurrent uncontrolled diseases
* Patients with malignant pleural or pericardial effusion.
* Previous treatments (radiotherapy treatment to the primary site, chemotherapy or treatment with tyrosine kinase inhibitor.)
* Pregnant or lactating women.
* Intercurrent malignant diseases, except basal cell carcinoma in skin inactive, carcinoma in situ of the cervix, when completely resected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-06; Primary Completion 2018-08 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of diagnosis until the date of death from any cause, assessed up to 100 months
  Time to event as calculated from confirmed histopathological diagnosis of NSCLC up until death or last follow up.

SECONDARY OUTCOMES:
Progression-free survival | From date of treatment start until the date of documented radiological (CT) progression, or date of death from any cause, whichever came first, assessed up to 100 months.
  Time to event as calculated from first-line therapy start (any therapy) until documented radiological progression as assessed by PET-CT using RECIST 1.1 criteria.
Complete metabolic response by PET-CT | From date of administration of first-line therapy (any therapy) until the date of metabolic progression as assessed by FDG PET-CT, date of death from any cause, whichever came first, assessed up to 100 months
  No evidence of metabolic activity by FDG PET-CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD, Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffioen GH, Toguri D, Dahele M, Warner A, de Haan PF, Rodrigues GB, Slotman BJ, Yaremko BP, Senan S, Palma DA. Radical treatment of synchronous oligometastatic non-small cell lung carcinoma (NSCLC): patient outcomes and prognostic factors. Lung Cancer. 2013 Oct;82(1):95-102. doi: 10.1016/j.lungcan.2013.07.023. Epub 2013 Aug 6. PMID 23973202
- [Background] De Ruysscher D, Wanders R, van Baardwijk A, Dingemans AM, Reymen B, Houben R, Bootsma G, Pitz C, van Eijsden L, Geraedts W, Baumert BG, Lambin P. Radical treatment of non-small-cell lung cancer patients with synchronous oligometastases: long-term results of a prospective phase II trial (Nct01282450). J Thorac Oncol. 2012 Oct;7(10):1547-55. doi: 10.1097/JTO.0b013e318262caf6. PMID 22982655
- [Background] Collen C, Christian N, Schallier D, Meysman M, Duchateau M, Storme G, De Ridder M. Phase II study of stereotactic body radiotherapy to primary tumor and metastatic locations in oligometastatic nonsmall-cell lung cancer patients. Ann Oncol. 2014 Oct;25(10):1954-1959. doi: 10.1093/annonc/mdu370. Epub 2014 Aug 11. PMID 25114022
- [Background] Ashworth A, Rodrigues G, Boldt G, Palma D. Is there an oligometastatic state in non-small cell lung cancer? A systematic review of the literature. Lung Cancer. 2013 Nov;82(2):197-203. doi: 10.1016/j.lungcan.2013.07.026. Epub 2013 Aug 20. PMID 24051084
- [Derived] Arrieta O, Barron F, Maldonado F, Cabrera L, Corona-Cruz JF, Blake M, Ramirez-Tirado LA, Zatarain-Barron ZL, Cardona AF, Garcia O, Aren O, De la Garza J. Radical consolidative treatment provides a clinical benefit and long-term survival in patients with synchronous oligometastatic non-small cell lung cancer: A phase II study. Lung Cancer. 2019 Apr;130:67-75. doi: 10.1016/j.lungcan.2019.02.006. Epub 2019 Feb 7. PMID 30885354